CLINICAL TRIAL: NCT07309237
Title: Spinning-Based High-Intensity Interval Training Induces Greater Cardiopulmonary Adaptations Than Continuous Training in Sedentary College Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fooyin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 113-233
Record Dates: First submitted 2025-11-21; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2024-08

CONDITIONS: Sedentary Lifestlye; Male

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high-intense interval training (Active Comparator): Performed repeated high-intensity bouts at 75-80% of VO₂ reserve, interspersed with active recovery at 60-65% of VO₂ reserve, using a spinning bike.
  Interventions: Behavioral: high intense interval training
- moderate-intensity continuous training (Placebo Comparator): At approximately 70% of VO₂ reserve, using a spinning bike.
  Interventions: Behavioral: moderate intense continue training; Behavioral: Control
- control group (No Intervention): did not perform any exercise training

INTERVENTIONS:
Behavioral: high intense interval training — performed repeated high-intensity bouts at 75-80% of VO₂ reserve, interspersed with active recovery at 60-65% of VO₂ reserve, using a spinning bike
  Arms: high-intense interval training
Behavioral: moderate intense continue training — continuously at approximately 70% of VO₂ reserve, using spinning bike
  Arms: moderate-intensity continuous training
Behavioral: Control — did not perform any exercise training
  Arms: moderate-intensity continuous training

SUMMARY:
In recent years, fitness concepts have continuously evolved, with many seeking to improve and enhance their physical condition through exercise to achieve better athletic performance. Aerobic exercise not only increases lipid utilization but also boosts athletic performance. Consequently, various aerobic exercise equipment has become increasingly popular in the market. Due to the pandemic's impact in recent years, people have rarely ventured outdoors, making indoor exercise equipment increasingly popular for home workouts. Spinning has emerged as a widely adopted new fitness activity, accessible to all genders and ages. Many gyms even offer specialized spinning classes with variations in speed and resistance. However, past literature has predominantly focused on continuous-intensity spinning interventions, which do not reflect the diverse training variations found in actual spinning classes. Therefore, this study aims to investigate the effects of incorporating high-intensity interval training (HIIT) into spinning on cardiorespiratory fitness.

ELIGIBILITY:
Inclusion Criteria:

* no regular exercise training in the past six months
* ability to safely perform high-intensity cycling exercise

Exclusion Criteria:

* musculoskeletal limitations that prevented cycling exercise
* recent infection
* known cardiopulmonary disease or medical history affecting cardiovascular or respiratory function
* smoking
* use of medications that may influence cardiopulmonary responses to exercise
* other contraindications to exercise testing according to the American College of Sports Medicine (ACSM) guidelines

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary fitness | Before intervention and the end of intervention at 6 weeks
  VO2max (ml/kg/mL)
Baseline anthropometric of the participants | Before intervention and the end of intervention at 6 weeks
  Age (yr)
Cardiopulmonary fitness | Before intervention and the end of intervention at 6 weeks
  VEmax (L/min)
Cardiopulmonary fitness | Before intervention and the end of intervention at 6 weeks
  maximal workload (W)
Cardiopulmonary fitness | Before intervention and the end of intervention at 6 weeks
  AT% (%VO₂max)
Cardiopulmonary fitness | Before intervention and the end of intervention at 6 weeks
  Resting O₂ pulse (mL·beat-¹)
Cardiopulmonary fitness | Before intervention and the end of intervention at 6 weeks
  Max O₂ pulse (mL·beat-¹)
Cardiopulmonary fitness | Before intervention and the end of intervention at 6 weeks
  MIP (cmH2O)
Cardiopulmonary fitness | Before intervention and the end of intervention at 6 weeks
  MEP (cmH2O)
Baseline anthropometric of the participants | Before intervention and the end of intervention at 6 weeks
  Height (cm)
Baseline anthropometric of the participants | Before intervention and the end of intervention at 6 weeks
  Weight (kg)
Baseline anthropometric of the participants | Before intervention and the end of intervention at 6 weeks
  BMI (kg/m²)

SECONDARY OUTCOMES:
Lung function | Before intervention and the end of intervention at 6 weeks
  FEV1 (L)
Lung functionWeight | Before intervention and the end of intervention at 6 weeks
  FVC (L)
Lung function | Before intervention and the end of intervention at 6 weeks
  FEV₁/FVC (%)
Lung function | Before intervention and the end of intervention at 6 weeks
  FEF25-75% (L·s-¹)
Lung function | Before intervention and the end of intervention at 6 weeks
  PEF (L·min-¹)
Lung function | Before intervention and the end of intervention at 6 weeks
  MVV (L·min-¹)
Lung function | Before intervention and the end of intervention at 6 weeks
  Breathing reserve (%)
Lung function | Before intervention and the end of intervention at 6 weeks
  Dynamic Index (DI%)

CONTACTS AND LOCATIONS:
Locations (1):
- No. 151, Jinxue Rd., Kaohsiung City, Daliao, Taiwan

IPD SHARING:
Plan to Share IPD: No